CLINICAL TRIAL: NCT05163509
Title: A Prospective, Phase II Study of MR-Linac Guided Adaptive Radiotherapy for Inoperable Mediastinal Tumor
Brief Title: MR-linac Guided Adaptive Radiotherapy for Inoperable Mediastinal Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1078
Record Dates: First submitted 2021-12-15; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Mediastinal Tumor
Keywords: Mediastinal Tumor; MR-Linac; Radiotherapy
MeSH Terms: conditions — Mediastinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-Linac Guided Adaptive Radiotherapy (Experimental): Patients will receive Adaptive Radiotherapy on the MR-Linac treatment machine.
  Interventions: Combination Product: Unity-based MR-Linac guided Radiotherapy

INTERVENTIONS:
Combination Product: Unity-based MR-Linac guided Radiotherapy — The radiotherapy was delivered using the Unity-based MR-Linac treatment machine.

SUMMARY:
This Phase II study is to determine the efficacy and safety of MR-Linac Guided Radiotherapy in patients with inoperable mediastinal tumors.

DETAILED DESCRIPTION:
This Phase II study is to determine the efficacy and safety of MR-Linac Guided Radiotherapy in patients with inoperable mediastinal tumors.

Patients will receive radiotherapy on the MR-Linac treatment machine. The primary end point is 2-year local-recurrence free survival. The secondary end points are objective response rate, 2-y PFS, 2-y OS, safety of treatment, dose coverage of targets and dose to normal organs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Histologically or cytologically confirmed mediastinal cancer
* Patients with inoperable mediastinal lesions
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Normal function of organs and bone marrow within 14 days: Total bilirubin 1.5 times or less the upper limits of normal (ULN); AST and ALT 1.5 times or less the ULN; absolute neutrophil count≥ 500 cells/mm3; creatinine clearance rate(CCR) ≥45 mL/min; Platelet count≥50,000 cells/mm3; international normalized ratio(INR) ≤1.5#Prothrombin Time (PT)≤ 1.5 × ULN
* Informed-consent

Exclusion Criteria:

* Patients with contraindications for MRI
* Previous radiotherapy or excision for mediastinal tumor
* The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava)
* A cavity over 2cm in diameter of primary tumor or metastasis Bleeding tendency or coagulation disorder
* Hemoptysis (1/2 teaspoon blood/day) happened within 1 month
* The use of full-dose anticoagulation within the past 1 month
* Severe vascular disease occurred within 6 months
* Gastrointestinal fistula, perforation or abdominal abscess occurred within 6 months
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg)
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours
* Urine protein 3-4+, or 24h urine protein quantitative >1g
* Severe uncontrolled disease
* Uncontrollable seizure or psychotic patients without self-control ability
* Women in pregnancy, lactation period
* Other not suitable conditions determined by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Local-recurrence free survival | 2 years

SECONDARY OUTCOMES:
Objective response rate | 2 months
Progression-free survival | 2 years
Overall survival | 2 years
Rate of patients with treatment-related adverse events evaluated by CTCAE v5.0 | 2 months
Dose coverage to targets and normal organs | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kunitoh H, Tamura T, Shibata T, Takeda K, Katakami N, Nakagawa K, Yokoyama A, Nishiwaki Y, Noda K, Watanabe K, Saijo N; JCOG Lung Cancer Study Group. A phase II trial of dose-dense chemotherapy, followed by surgical resection and/or thoracic radiotherapy, in locally advanced thymoma: report of a Japan Clinical Oncology Group trial (JCOG 9606). Br J Cancer. 2010 Jun 29;103(1):6-11. doi: 10.1038/sj.bjc.6605731. Epub 2010 Jun 15. PMID 20551960
- [Background] Jaffray DA, Siewerdsen JH, Wong JW, Martinez AA. Flat-panel cone-beam computed tomography for image-guided radiation therapy. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1337-49. doi: 10.1016/s0360-3016(02)02884-5. PMID 12128137
- [Background] Lagendijk JJ, Raaymakers BW, Van den Berg CA, Moerland MA, Philippens ME, van Vulpen M. MR guidance in radiotherapy. Phys Med Biol. 2014 Nov 7;59(21):R349-69. doi: 10.1088/0031-9155/59/21/R349. Epub 2014 Oct 16. No abstract available. PMID 25322150
- [Background] Khoo VS, Joon DL. New developments in MRI for target volume delineation in radiotherapy. Br J Radiol. 2006 Sep;79 Spec No 1:S2-15. doi: 10.1259/bjr/41321492. PMID 16980682
- [Background] Raaymakers BW, Lagendijk JJ, Overweg J, Kok JG, Raaijmakers AJ, Kerkhof EM, van der Put RW, Meijsing I, Crijns SP, Benedosso F, van Vulpen M, de Graaff CH, Allen J, Brown KJ. Integrating a 1.5 T MRI scanner with a 6 MV accelerator: proof of concept. Phys Med Biol. 2009 Jun 21;54(12):N229-37. doi: 10.1088/0031-9155/54/12/N01. Epub 2009 May 19. PMID 19451689
- [Background] Stemkens B, Tijssen RH, de Senneville BD, Lagendijk JJ, van den Berg CA. Image-driven, model-based 3D abdominal motion estimation for MR-guided radiotherapy. Phys Med Biol. 2016 Jul 21;61(14):5335-55. doi: 10.1088/0031-9155/61/14/5335. Epub 2016 Jun 30. PMID 27362636
- [Background] Dietz B, Yip E, Yun J, Fallone BG, Wachowicz K. Real-time dynamic MR image reconstruction using compressed sensing and principal component analysis (CS-PCA): Demonstration in lung tumor tracking. Med Phys. 2017 Aug;44(8):3978-3989. doi: 10.1002/mp.12354. Epub 2017 Jun 28. PMID 28543069
- [Background] Glitzner M, Crijns SP, de Senneville BD, Kontaxis C, Prins FM, Lagendijk JJ, Raaymakers BW. On-line MR imaging for dose validation of abdominal radiotherapy. Phys Med Biol. 2015 Nov 21;60(22):8869-83. doi: 10.1088/0031-9155/60/22/8869. Epub 2015 Nov 4. PMID 26531846
- [Background] Kontaxis C, Bol GH, Stemkens B, Glitzner M, Prins FM, Kerkmeijer LGW, Lagendijk JJW, Raaymakers BW. Towards fast online intrafraction replanning for free-breathing stereotactic body radiation therapy with the MR-linac. Phys Med Biol. 2017 Aug 21;62(18):7233-7248. doi: 10.1088/1361-6560/aa82ae. PMID 28749375
- [Background] Raaymakers BW, Jurgenliemk-Schulz IM, Bol GH, Glitzner M, Kotte ANTJ, van Asselen B, de Boer JCJ, Bluemink JJ, Hackett SL, Moerland MA, Woodings SJ, Wolthaus JWH, van Zijp HM, Philippens MEP, Tijssen R, Kok JGM, de Groot-van Breugel EN, Kiekebosch I, Meijers LTC, Nomden CN, Sikkes GG, Doornaert PAH, Eppinga WSC, Kasperts N, Kerkmeijer LGW, Tersteeg JHA, Brown KJ, Pais B, Woodhead P, Lagendijk JJW. First patients treated with a 1.5 T MRI-Linac: clinical proof of concept of a high-precision, high-field MRI guided radiotherapy treatment. Phys Med Biol. 2017 Nov 14;62(23):L41-L50. doi: 10.1088/1361-6560/aa9517. PMID 29135471